CLINICAL TRIAL: NCT02251405
Title: Behaviour Intervention to Decrease Melamine Exposure
Acronym: Bidme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ming-Tsang Wu (Other)
Responsible Party: Sponsor-Investigator, Ming-Tsang Wu, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Organization: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KMU-DT103004; KMU-DT103004 (Other: Kaohsiung Medical University Hospital)
Record Dates: First submitted 2014-08-08; First posted 2014-09-29 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Subjects
Keywords: Melamine; Melamine tableware

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One big bag, no stainless container (Placebo Comparator): No stainless container
  Interventions: Behavioral: One bag, stainless container
- One big bag with two stainless containers (Active Comparator): Two stainless containers
  Interventions: Behavioral: One bag, stainless container

INTERVENTIONS:
Behavioral: One bag, stainless container

SUMMARY:
One source of melamine exposure in the modern life is from the use of melamine tableware. This study examines whether the use of stainless steel containers can decrease melamine exposure in the daily life. The investigators hypothesize that, compared to those without use of stainless steel containers, university student volunteers with use of stainless steel containers excrete significantly lower melamine levels in urine.

DETAILED DESCRIPTION:
Study subjects:

Two tiers:

1. Recruit 88 student volunteers from two university buildings and collect their morning one-spot urine specimens for 3 consecutive days (44 students in each building (Building A and Building B)
2. Select appropriate study subjects with high excretion of urinary melamine and with consuming melamine tableware containing hot water or hot soup by questionnaire in the past 3 days for intervention.

Study protocol:

This is a cluster randomized crossover intervention. We will conduct this study for 9 days and each experimental step lasts for 3 days. We randomly assign one building with 8 appropriate study subjects to a serial of control-intervention-intervention steps and another building with also 8 appropriate study subjects to a serial of control-control-intervention steps. Intervention step means study subjects will carry one big bag containing two stainless containers, one stainless spoon, and one stainless chopstick and use them for each meal during the trial (Some subjects will need to take pictures randomly and email back before the meal). Control means study subjects will carry one big bag without those stainless container, spoon, and chopstick and only use the containers provided by vendors for each meal during the trial (Some subjects will need to take pictures randomly and email back before the meal to check their adherence). Collect 24-hr urine samples for 9 days for melamine levels.

Inclusion criteria: 20-30 healthy students Exclusion criteria: Subjects with cancer, hypertension, diabetes, chronic hepatic or renal diseases, including urinary tract infection, or renal stones; Family history of renal stones; Body weight less than 50 kg.

ELIGIBILITY:
Inclusion Criteria:

* 20-30-yrs healthy students

Exclusion Criteria:

* Subjects with cancer, hypertension, diabetes, chronic hepatic or renal diseases, renal stones;
* Family history of renal stones;
* Body weight less than 50 kg.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Decrease melamine excretion | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tsang Wu, MD, ScD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan